CLINICAL TRIAL: NCT07208227
Title: In-use Tolerance and Efficacy Study Under Dermatological and Ophthalmological Controls - Face Cream, RV4983A - LA3365
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4983A20210135
Record Dates: First submitted 2025-09-15; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Sensitive Skin; Deep Wrinkles
Keywords: open trial; antiaging cosmetic cream

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group
  Interventions: Other: Face Cream RV4983A LA3365

INTERVENTIONS:
Other: Face Cream RV4983A LA3365 — Cosmetic face cream product applied once a day on face, neck and neckline.

SUMMARY:
Tolerance and efficacy study of an anti aging cream on 44 subjects aged between 45 and 65 years, with sensitive skin and deep wrinkles. This study is conducted as a national, monocentric, non-randomized open trial.

Planning of the visits:

* Visit 1: Inclusion (Day 1)
* Visit 2: Intermediate visit (Day 29), a window of +48 hours is allowed
* Visit 3: End of study (Day 57), a window of +72 hours is allowed The maximum duration of participation for a subject is 60 days.

ELIGIBILITY:
INCLUSION CRITERIA

Criteria related to the population:

* female
* aged between 45 and 65 years included
* phototype: I to III
* skin type: oily, combination, normal, dry, very dry
* 100% of subjects with sensitive skin on the face
* 100% of subjects with deep wrinkles on the face
* 100% of subjects with sagging skin on the face
* 100% of subjects with dull and uneven complexion
* subjects must be registered with health social security or health social insurance
* having signed their written Informed Consent form (ICF) for their participation in the study and a photograph authorization
* certifying the truth of the personal information declared to the Investigator
* able to understand the language used in the investigation centre and the information given
* able to comply with the protocol and follow protocol's constraints and specific requirements
* a maximum of 20% of subjects being lens wearers will be included in the study
* subject agree to not expose herself to sunlight or UV during the study and if necessary, provide sun protection

Criteria related to subject's health:

* considered "healthy subject" by the Investigator
* women of childbearing potential committing themselves to use effective contraceptive method throughout the study and for at least 3 months before the inclusion visit

NON INCLUSION CRITERIA

Criteria related to the population:

* having participated in another clinical trial within the week before the inclusion visit and for a longer period if required in the Investigator's opinion
* taking part or planning to participate in another clinical trial during the study in the same or another investigation centre
* deprived of freedom by administrative or legal decision or under guardianship
* not able to be contacted in case of emergency
* admitted in a sanitary or social facilities o planning an hospitalization during the study
* belonging to the staff of the investigation centre

Criteria related to subject's health:

* breastfeeding, pregnant (for the women of childbearing potential)
* having a dermatological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* having an ophthalmological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* having personal medical history liable to interfere with the study data for the subject (especially characterized cosmetic hyperreactivity) or incompatible with the study requirements (except if this population is required by the Sponsor i.e atopic dermatitis)
* having history of abnormal reactions from exposure to sunlight
* having taken any previous treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements
* being under any treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements

Criteria related to investigational product application areas:

* having had any surgery, chemical or significant invasive dermo-treatment on the experimental area considered by the Investigator liable to interfere with the study data, before the inclusion visit or foreseeing it for the duration of the study
* having applied a skincare or make up product on the study areas the day of the inclusion visit. The usual cleanser is allowed.
* having received, on the study areas, artificial UV exposure or excessive exposure to natural sunlight within the 1 month before the inclusion visit

Criteria related to the COVID-19 pandemic:

* Subject who was abroad in a country with a higher incidence rate of Covid-19 than Poland, within 14 days before the beginning of the study
* Subject presenting following symptoms: cough, shortness of breath, elevated body temperature - equal or above 37,5°C
* Subject who had contact with any person infected with COVID-19 within 10 days before the beginning of the study
* Subject who is currently during home quarantine recommended by the Sanitary Inspection

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the investigation centre's panel. They will be selected on the basis of inclusion and non-inclusion criteria specific to the study. They will be definitely included in the study after a specific interview and a clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Global tolerance assessment | At the end of the study, after Last Patient Out, (after Day 57)
  Global tolerance is assessed on the "tolerance population" which includes all the subjects who applied at least once investigational product.
  Global assessment of the dermatological and ophthalmological tolerance is done by the investigator. This assessment allows for attribution of one of the 5 levels : excellent, very good, good, moderate, bad.

SECONDARY OUTCOMES:
Ra parameter to evaluate smoothing/anti-wrinkle effect | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Ra= Average roughness Ra is the arithmetic mean of the absolute values (without differentiation between peaks and valleys) of the heights of the profile length.
  Measured by 3D PRIMOS-CR SYSTEM
Rz parameter to evaluate smoothing/anti-wrinkle effect | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Rz= Average height of the roughness= Average relief Rz is the average of 5 single roughness depths, measured within the section ln. The single roughness depth is the difference from the highest profile peak to the deepest profile valley within a single measurement section.
  Measured by 3D PRIMOS-CR SYSTEM
Rt parameter to evaluate smoothing/anti-wrinkle effect | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Rt= Maximum height of the roughness profile= maximum relief amplitude Rt is the height difference from the highest peak to the deepest valley within the total measurement section Measured by 3D PRIMOS-CR SYSTEM
Clinical scoring of the visibility of crow's feet wrinkles | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by the investigator according to the BAZIN scale (7-point scale, from 0 to 6)
Clinical scoring of the Smoothness of the skin | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by the investigator on a 11-point scale (0 = rough skin, 10 = very smooth skin)
Clinical scoring of the Firmness of the skin | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by the investigator on a 11-point scale (0 = sagged skin, 10 = very firm skin)
Clinical scoring of the Skin plumpness | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by the investigator on a 11-point scale (0 = thin and not replumped skin, 10 = very replumped skin)
Clinical scoring of Radiance/ Luminosity based on photographs | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by three jury assessors who assess the parameter on unstructured scales (corresponding to scores from 0 to 10, 0= dull, 10= radiant/luminous) based on photographs taken by Colorface
Clinical scoring of Skin brightness based on photographs | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by three jury assessors who assess the parameter on unstructured scales (corresponding to scores from 0 to 10, 0= not bright at all, 10= very bright) based on photographs taken by Colorface
Clinical scoring of homogeneity of skin tone based on photographs | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by three jury assessors who assess the parameter on unstructured scales (corresponding to scores from 0 to 10, 0= not even at all, 10= very even) based on photographs taken by Colorface
Clinical scoring of homogeneity of skin texture based on photographs | Visit 1 (Day 1, before investigational product application), Visit 2 (Day 29) and Visit 3 (Day 57).
  Assessed by three jury assessors who assess the parameter on unstructured scales (corresponding to scores from 0 to 10, 0= coarse, 10= fine) based on photographs taken by Colorface

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Poland Sp. z o. o, Gdansk, Poland, Poland